CLINICAL TRIAL: NCT07023146
Title: Adaptations Due to Different Intensities of Power Training on Neuromuscular Performance, Muscle Thickness and Functional Capacity in Elderly People: A Randomized Clinical Trial
Brief Title: Effects of Different Power Training Intensities in Older Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Antenor Barbosa Calandrini de Azevedo, Doctor Student, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 85503024.6.0000.5347
Record Dates: First submitted 2025-05-23; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Investigating the Effects of Power Training in the Elderly
Keywords: Aging; resistance training; functional capacity; muscle strength; muscle hypertrophy
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: The methodological procedures of this project will be carried out at the UFRGS facilities, on the campus of the School of Physical Education, Physiotherapy and Dance (ESEFID) and at LAPEX. After two weeks of familiarization, in order to guarantee the reproducibility and reliability of the methodological procedures, the participants will be randomized electronically (randomizer.org.br) to perform low to moderate intensity (PTLM; 40-60% of 1-repetition maximum [1RM]) and moderate to high intensity (PTMH; 65-80% of 1RM).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low to moderate intensity (PTLM; 40-60% of 1-repetition maximum [1RM]) (Active Comparator): Power training performed at maximum velocity in the concentric phase with lower to moderate intensity
  Interventions: Device: low to moderate intensity (PTLM; 40-60% of 1-repetition maximum [1RM])
- Moderate to high intensity (PTMH; 65-80% % of 1-repetition maximum [1RM]) (Active Comparator): Power training performed at maximum velocity in the concentric phase with moderate to high intensity
  Interventions: Device: Moderate to high intensity (PTMH; 65-80% of 1-repetition maximum [1RM]) )

INTERVENTIONS:
Device: Moderate to high intensity (PTMH; 65-80% of 1-repetition maximum [1RM]) ) — Power training performed at maximum velocity in the concentric phase with moderate to high intensity
  Other Names: PTMH; Linear Encoder; Load Cell; 1-Repetition Maximum (1RM); Ultrasound
  Arms: Moderate to high intensity (PTMH; 65-80% % of 1-repetition maximum [1RM])
Device: low to moderate intensity (PTLM; 40-60% of 1-repetition maximum [1RM]) — Power training performed at maximum velocity in the concentric phase with lower to moderate intensity
  Other Names: PTLM; Linear Encoder; 1-Repetition Maximum (1RM); Ultrasound; Load Cell
  Arms: Low to moderate intensity (PTLM; 40-60% of 1-repetition maximum [1RM])

SUMMARY:
Power (strength × velocity) is a crucial component for maintaining independence during aging. Therefore, investigating interventions aimed at improving this physical capacity is essential for this population. The aim of this study is to examine the effects of power training (PT) performed at low to moderate intensity (PTLM; 40-60% of 1-repetition maximum [1RM]) and moderate to high intensity (PTMH; 65-80% of 1RM) on muscle power, kinematic gait parameters, strength, muscle thickness, and functional performance in older adults. Participants will be randomly assigned to perform PTLM and PTMH. Data collection will occur before and after familiarization, as well as at weeks 8 and 16 of the training programs. Participants will undergo a series of tests in the following sequence: 1) muscle thickness and 1RM test; 2) muscle power, maximum voluntary contraction, and rate of force development; 3) functional performance. The primary analyses will be conducted on an intention-to-treat basis, comparing the effects of the interventions and groups over time. Generalized Estimating Equations (GEE) will be used, considering the factors of group (2 levels) and time (3 levels). Paired comparisons will be assessed using the Bonferroni post-hoc test to identify significant differences between groups and time points. All tests will be performed using JASP software (version 0.16.4.0), with statistical significance set at p < 0.05 for all analyses.

ELIGIBILITY:
Inclusion criteria:

* Age 60 years or older
* No participation in regular and systematic resistance training in the last three months
* No absolute or relative contraindications to exercise
* No musculoskeletal injuries that could interfere with training and assessments

Exclusion criteria:

* Use of steroids, nutritional supplements, or ergogenic substances
* Failure to complete all study phases
* Failure to complete more than 80% of the training sessions (32 sessions)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-12-11 (Estimated); Study Completion 2025-12-11 (Estimated)

PRIMARY OUTCOMES:
Muscle Power | Pre- and post-intervention (16 weeks of training)
  The power output during strength exercises is assessed using an encoder linear at two different intensities: 30% and 70% of 1RM in leg extension and leg press 45. Power output is the ability to generate force quickly and is a key measure of explosive strength. These tests are performed using different resistance levels to assess power across a range of intensities.
  Measurement Tool: Encoder linear (linear encoder or velocity-based device)
  Scale: Power output in watts (W)
  Higher scores indicate better power performance at each intensity.
Muscle Strength | Pre- and post-intervention (16 weeks of training)
  Muscle strength is the ability of a muscle or muscle group to generate force against resistance. It reflects the maximum force that can be produced in a single effort and is essential for daily activities and overall physical function. One Repetition Maximum (1RM) is used to quantify maximal strength.
  Measurement Tool: 1RM testing
  Scale: 1RM (measured in kg)
  Higher scores indicate better strength performance.
Rate of Force Development | Pre- and post-intervention (16 weeks of training)
  Rate of force development refers to the speed at which force is generated by a muscle or muscle group. It is a critical measure of neuromuscular performance, especially in activities that require explosive strength or rapid reactions. RFD is measured during maximal voluntary contractions.
  Measurement Tool: Load Cell
  Scale: Measured in Newtons per second (N/s)
  Higher scores indicate better neuromuscular performance.

SECONDARY OUTCOMES:
Functional Capacity | Pre- and post-intervention (16 weeks of training)
  Functional capacity refers to an individual's ability to perform activities required for daily living, such as walking, climbing stairs, or carrying objects. It reflects overall physical function and is often used to assess health status, particularly in older adults or clinical populations. The following tests were selected to assess functional capacity:
  Stair Climbing Test Scale: Total time to climb and descend a predetermined number of stairs. Shorter time indicates better performance. Timed Up and Go (TUG) Scale: Total time in seconds. Shorter time indicates better mobility and agility. 6-Meter Walk Speed Test Scale: Total time to walk 6 meters (seconds). Shorter time indicates faster walking speed. Sit-to-Stand Test (5 times) Scale: Total time to complete the 5 repetitions. Shorter time indicates better muscle strength and functional capacity.
Muscle hypertrophy | Pre- and post-intervention (16 weeks of training)
  Muscle thickness is an indicator of muscle size and hypertrophy. It reflects the structural adaptations that occur in response to training. Ultrasound is used to measure the thickness of muscles such as the quadriceps, biceps, and triceps.
  Measurement Tool: Ultrasound imaging
  Scale: Muscle thickness in millimeters (mm)
  Higher scores indicate greater muscle hypertrophy.
Cognitive Capacity | Pre- and post-intervention (16 weeks of training)
  The Montreal Cognitive Assessment (MoCA) is a brief screening tool used to assess cognitive function. It evaluates multiple cognitive domains, including memory, attention, language, and executive functions. It is commonly used to assess cognitive decline or impairments.
  Measurement Tool: MoCA test
  Scale: MoCA score ranges from 0 to 30, with higher scores indicating better cognitive function.
  Higher scores indicate better cognitive function.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio Grande do Sul (UFRGS), Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinikorena I, Martinez-Ramirez A, Gomez M, Lecumberri P, Casas-Herrero A, Cadore EL, Millor N, Zambom-Ferraresi F, Idoate F, Izquierdo M. Gait Variability Related to Muscle Quality and Muscle Power Output in Frail Nonagenarian Older Adults. J Am Med Dir Assoc. 2016 Feb;17(2):162-7. doi: 10.1016/j.jamda.2015.09.015. Epub 2015 Nov 11. PMID 26577625
- [Background] Mc Dermott EJ, Balshaw TG, Brooke-Wavell K, Maden-Wilkinson TM, Folland JP. Fast and ballistic contractions involve greater neuromuscular power production in older adults during resistance exercise. Eur J Appl Physiol. 2022 Jul;122(7):1639-1655. doi: 10.1007/s00421-022-04947-x. Epub 2022 Apr 16. PMID 35429294
- [Background] Bandeira-Guimaraes M, Blanco-Rambo E, Vieira AF, Saez de Asteasu ML, Pinto RS, Izquierdo M, Cadore EL. Chronic Effects of Different Intensities of Power Training on Neuromuscular Parameters in Older People: A Systematic Review with Meta-analysis. Sports Med Open. 2023 Oct 24;9(1):98. doi: 10.1186/s40798-023-00646-9. PMID 37874417
- [Background] de Vos NJ, Singh NA, Ross DA, Stavrinos TM, Orr R, Fiatarone Singh MA. Optimal load for increasing muscle power during explosive resistance training in older adults. J Gerontol A Biol Sci Med Sci. 2005 May;60(5):638-47. doi: 10.1093/gerona/60.5.638. PMID 15972618
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37874417/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15972618/